CLINICAL TRIAL: NCT02021227
Title: Effects of Chair Sitting Exercise Intervention on Weaning From Mechanical Ventilation and Mortality of Critically Ill Patients With Acute Respiratory Failure: a Randomised Controlled Trial.
Brief Title: Early Chair Sitting Exercise in Mechanically Ventilated Critically Ill Patients
Acronym: RehabVent
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sufficient enrollment
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9231
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Chronic Respiratory Failure With Acute Decompensation Requiring Mechanical Ventilation for More Than 48 Hours
Keywords: Acute respiratory failure; Mechanical ventilation; Rehabilitation; Exercise chair sitting; Weaning; Chronic respiratory failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard group (No Intervention)
- Chair sitting group (Other)
  Interventions: Procedure: Early chair sitting exercise

INTERVENTIONS:
Procedure: Early chair sitting exercise — A chair sitting exercise will be done at least once a day and for > 1 hour
  Arms: Chair sitting group

SUMMARY:
The occurrence of an acute respiratory failure necessitates mostly admission to ICU and mechanical ventilation (MV). Rapid and safe discontinuation of MV should be the objective for the majority of patients. Many reasons may contribute to weaning, extubation failure and prolongation of MV. Critical illness myopathy, induced by immobilisation and prolonged MV, may represent a main factor and early rehabilitation may reverse these conditions and improve the success of weaning from MV.The objective of this study is to evaluate the effect of an early chair sitting (while the patient is awake but still mechanically ventilated) on weaning from mechanical ventilation and ICU mortality.

Methods: Chronic respiratory failure patients with an acute decompensation and requiring MV for more than 48 hours will be randomized to 2 groups at the initiation of weaning schedule: the studied group (20 patients): chair-sitting group will be transferred from bed to arm chair for at least 1 hour and once a day; the control group will stay in bed until extubation. Ventilator free days, extubation failure, nosocomial infections, ICU mortality, ICU length of stay are assessed and compared between groups. Expected results: Early chair sitting would decrease MV duration, number of extubation failure, nosocomial infections and ICU mortality. Feasibility and safety of this intervention will also be evaluated and also the related work load.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure
* Requiring mechanical ventilation for more than 48 h
* Informed consent

Exclusion Criteria:

* Body mass index > 40 kg/m2
* Severe neuropathy
* Hemodynamic instability, acute cor pulmonary embolism, acute myocardial ischemia/necrosis, hypoxemia
* Deep sedation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Weaning from mechanical ventilation, mortality | day 28

SECONDARY OUTCOMES:
ICU length of stay | day 28
Extubation success | day 28
  success or failure
Nosocomial infections | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Kada KLOUCHE, MD PhD, Principal Investigator — Hopital de Montpellier
Locations (1):
- Lapeyronie University Hospital, Intensive Care Department, Montpellier, France

REFERENCES:
- [Result] Canaud B, Formet C, Raynal N, Amigues L, Klouche K, Leray-Moragues H, Beraud JJ. Vascular access for extracorporeal renal replacement therapy in the intensive care unit. Contrib Nephrol. 2004;144:291-307. doi: 10.1159/000078897. No abstract available. PMID 15264418